CLINICAL TRIAL: NCT00593268
Title: Biological Markers of Vasospasm in Cerebral Spinal Fluid and Blood in Patients With Subarachnoid Hemorrhage
Brief Title: Evaluation of Cerebral Spinal Fluid and Blood in Patients With Subarachnoid Hemorrhage
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Reid Thompson, Professor of Neurological Surgery, Vanderbilt University Medical Center
Other Study IDs: 031084
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — cerebrospinal fluid and blood
Oversight: Data Monitoring Committee: No

SUMMARY:
In this project we are collecting cerebrospinal fluid and blood from patients at Vanderbilt Medical Center who have a subarachnoid hemorrhage which has followed the rupture of a brain aneurysm. We then propose to study the cerebrospinal fluid using a novel microscopic laser directed mass spectrometric analysis (MALDI) available at Vanderbilt. The cerebrospinal fluid and blood will then be analysed for different biological markers, protein expression and gene expression. These markers will then be statistically correlated with clinical data including prediction of vasospasm, time to vasospasm and response to standard therapy.

DETAILED DESCRIPTION:
In this project we are collecting cerebrospinal fluid and blood from patients at Vanderbilt Medical Center who have a subarachnoid hemorrhage which has followed the rupture of a brain aneurysm. We then propose to study the cerebrospinal fluid using a novel microscopic laser directed mass spectrometric analysis (MALDI) available at Vanderbilt. The cerebrospinal fluid and blood will then be analysed for different biological markers, protein expression and gene expression. These markers will then be statistically correlated with clinical data including prediction of vasospasm, time to vasospasm and response to standard therapy.

The goal of this study is to determine cerebrospinal fluid and serum markers which will be predictive of vasospasm. This in turn may lead to improved outcomes in this population of patients.

The data will be compared to excess cerebrospinal fluid collected from patients who are undergoing lumbar puncture in the Neurology Clinic or excess cerebrospinal fluid from patients undergoing cranial surgery for other causes like tumor excision.

For patients enrolled in the study, cerebrospinal fluid will be collected by either lumbar puncture or external ventricular catheter. Specimens will be collected immediately pre-operatively if an external ventricular drain is in place or intraoperatively if an external ventricular drain is not present. We will also collect cerebrospinal fluid post operatively after placement of an external ventricular drain regularly from the excess cerebrospinal fluid that has been collected in the drainage bag. CSF will be collected in a serial fashion at multiple time points: immediately post operatively, during vasospasm and before the external ventricular drain is removed.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible to participate in this study are those that have a documented subarachnoid hemorrhage from a ruptured cerebral aneurysm or patients who have excess cerebrospinal fluid after a Lumbar Puncture or surgery for tumor resection.
* 18 years of age or older

Exclusion Criteria:

* Patients or family who are unable to understand the informed consent process will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 years of age or older
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2004-06; Primary Completion 2015-11 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
correlate biological markers of cerebral vasospasm with clinical outcomes | post hemorrhage
  Correlation of blood biological markers and clinical outcomes of cerebral vasospasm

CONTACTS AND LOCATIONS:
Overall Officials: Reid C. Thomspon, M.D., Principal Investigator — Vanderbilt University Medical Center, Department of Neurological Surgery
Locations (1):
- Vanderbilt University Medical Center, Department of Neurological Surgery, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided